CLINICAL TRIAL: NCT05710705
Title: Bioimpedance Measurement of Abdominal Free Flaps During Arterial and Venous Weaning in Breast Reconstruction
Acronym: MONITRANS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: PI2022_843_0040
Record Dates: First submitted 2022-12-08; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-12

CONDITIONS: Breast Reconstruction; Thrombosis, Venous; Bioimpedance Measurement Capacity
Keywords: breast reconstruction; Thrombosis, Venous; bioimpedance measurement capacity
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: portable prototype of bioimpedance measurement — The device will be installed during the patient's operation. It will be attached to the healthy skin of the flap (without wound or scar) by sterile glue. It will then be covered with a self-adhesive "tegaderm" type dressing. The wound will be isolated from the device with a hermetic silicone dressing of the "Mepilex" type, for example. There will therefore be no communication between the measuring device and the surgical wound.

SUMMARY:
As the occurrence of thrombosis in post surgery is rare, it seemed difficult to study only this one. This is why we decided to test the bioimpedance, temperature and green, red and infrared light absorption measurements of the prototype during the weaning of the flap during surgery. Indeed, during weaning the investigators voluntarily interrupt the arterial and venous flow to transfer the flap to the breast. This weaning corresponds to a thrombosis model.

The patients will benefit from an "improved" postoperative monitoring. Indeed, in addition to the classical clinical monitoring, they will benefit from an additional monitoring during 5 days thanks to the realization of an ultrasound of the flap which will be carried out every 6 hours the first 24 hours then every 12 hours.

This protocol is therefore a feasibility study for the collection of data of interest.

ELIGIBILITY:
Inclusion Criteria:

* Woman undergoing microsurgical breast reconstruction using a free abdominal flap
* Age greater than or equal to 18 years

Exclusion Criteria:

* Pregnant patient
* Patient with an active implantable device such as a pacemaker or an artificial heart
* Patient refusing to participate in the study
* Age less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast reconstruction
Enrollment: 10 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of impedence | one day
  Impedence measurement during episode of ischemia.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No